CLINICAL TRIAL: NCT02151981
Title: A Phase III, Open Label, Randomized Study of AZD9291 Versus Platinum-Based Doublet Chemotherapy for Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Whose Disease Has Progressed With Previous Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy and Whose Tumours Harbour a T790M Mutation Within the Epidermal Growth Factor Receptor Gene (AURA3).
Brief Title: AZD9291 (Osimertinib) Versus Platinum-Based Doublet-Chemotherapy in Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Acronym: AURA3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5160C00003; 2014-000594-39 (EudraCT Number)
Record Dates: First submitted 2014-05-15; First posted 2014-06-02 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Anticancer Treatment
Keywords: Advanced Non-Small Cell Lung Cancer; T790M Mutation Positive
MeSH Terms: interventions — Drug Therapy; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osimertinib (Experimental): Osimertinib 80 mg, orally, once daily
  Interventions: Drug: Chemotherapy; Drug: Cross-over to Osimertinib
- Platinum-based doublet chemotherapy (Active Comparator): pemetrexed 500mg/m2 + carboplatin AUC5 or pemetrexed 500mg/m2 + cisplatin 75mg/m2
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Randomization to either Osimertinib or platinum-based doublet-chemotherapy on Day 1 of every 21d cycle in a 2:1 (Osimertinib:platinum-based doublet-chemotherapy) ratio
  Other Names: Osimertinib; Platinum-based Doublet-Chemotherapy
Drug: Cross-over to Osimertinib — Once subjects on the platinum-based doublet chemotherapy arm are determined to have objective radiological progression according to RECIST 1.1 by the investigator and confirmed by independent central imaging review, they will be given the opportunity to begin treatment with Osimertinib 80mg, once daily. These subjects may continue treatment with Osimertinib even after disease progression, as long as they are continuing to show clinical benefit, as judged by the investigator.
  Subjects who stop platinum-based doublet chemotherapy for reasons other than objective disease progression according to RECIST 1.1 will not be eligible to cross-over to Osimertinib.
  Arms: Osimertinib

SUMMARY:
A Phase III, Open Label, Randomized Study of Osimertinib versus Platinum-Based Doublet Chemotherapy for Patients with Locally Advanced or Metastatic Non-Small Cell Lung Cancer whose Disease has Progressed with Previous Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy and whose Tumours harbour a T790M mutation within the Epidermal Growth Factor Receptor Gene

DETAILED DESCRIPTION:
This is a phase III, open label, randomized study assessing Osimertinib (80 mg, orally, once daily) versus platinum-based doublet chemotherapy (standard of care) in subjects with confirmed diagnosis of Epidermal Growth Factor Receptor (EGFR) mutation positive NSCLC, who have progressed following prior therapy with an approved Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) agent and whose tumours harbour a T790M mutation within the EGFR Gene. Subjects must be chemotherapy naive and must agree to provide a biopsy for central confirmation of T790 mutation status following confirmed disease progression on their first line EGFR-TKI treatment (e.g. erlotinib, gefitinib or afatinib). Suitable subjects will then be randomized to receive either Osimertinib (80mg orally, once daily) or platinum-based doublet chemotherapy (pemetrexed 500 mg/m2 + carboplatin area under the plasma concentration-time curve AUC 5 or pemetrexed 500 mg/m2 + cisplatin 75 mg/m2) on Day 1 of every 21-day cycle in a 2:1 (Osimertinib: platinum-based doublet chemotherapy) ratio. Once subjects on the platinum-based doublet chemotherapy arm are determined to have objective radiological progression according to RECIST 1.1 by the investigator and confirmed by independent central imaging review, they will be given the opportunity to begin treatment with Osimertinib 80mg, once daily. These subjects may continue treatment with Osimertinib even after disease progression, as long as they are continuing to show clinical benefit, as judged by the investigator. The primary objective of the study is to assess the efficacy of Osimertinib compared with platinum-based doublet chemotherapy by assessment of Progression Free Survival (PFS), using investigator assessments according to Response Evaluation Criteria in Solid Tumours (RECIST 1.1), as well as asensitivity analysis of Progression Free Survival using Blinded Independent Central Review (BICR).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically documented NSCLC.
* Locally advanced or metastatic NSCLC
* Radiological documentation of disease progression following 1st line EGFR TKI Treatment without any further treatment
* Eligible to receive treatment with the selected doublet-chemotherapy
* Central confirmation of T790M+ mutation status
* World Health Organization (WHO) performance status 0-1
* At least one lesion, not previously irradiated.

Exclusion Criteria:

* • Prior neo-adjuvant or adjuvant chemotherapy treatment within 6 months prior of starting 1st EGFR TKI treatment
* Treatment with more than one prior line of treatment for advanced NSCLC
* Treatment with an approved EGFR-TKI (e.g.,erlotinib, gefitinib, afatinib) within 8 days or approximately 5x half-life of the first dose of study treatment
* Any investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment
* Previous treatment with Osimertinib, or a 3rd generation EGFR TKI

For subjects who cross-over to Osimertinib:

* Once subjects on the platinum-based doublet chemotherapy arm are determined to have objective radiological progression according to RECIST 1.1 by the investigator and confirmed by independent central imaging review.
* At least 14 days since last dose of platinum-based doublet chemotherapy

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong General Hospital, Guangdong, 510030, China; Vassiliki A Papadimitrakopoulou, MD, Principal Investigator — The University of Texas/M.D. Anderson Cancer Center, Houston, Tx, USA
Locations (129):
- United States (21):
  - Research Site, Anaheim, California
  - Research Site, Orange, California
  - Research Site, Santa Rosa, California
  - Research Site, Norwalk, Connecticut
  - Research Site, Gainesville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Park Ridge, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Marrero, Louisiana
  - Research Site, Chevy Chase, Maryland
  - Research Site, Lebanon, New Hampshire
  - Research Site, Brick, New Jersey
  - Research Site, New York, New York
  - Research Site, Hershey, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Houston, Texas
  - Research Site, Lacey, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Milwaukee, Wisconsin
- Australia (5):
  - Research Site, Darlinghurst
  - Research Site, Heidelberg
  - Research Site, Kogarah
  - Research Site, Nedlands
  - Research Site, Woolloongabba
- Canada (6):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (12):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Nanchang
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Zhengzhou
- France (8):
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (6):
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Gerlingen
  - Research Site, Oldenburg
  - Research Site, Regensburg
  - Research Site, Würzburg
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Research Site, Budapest, Hungary
- Italy (5):
  - Research Site, Avellino
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Roma
- Japan (22):
  - Research Site, Akashi-shi
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hirakata-shi
  - Research Site, Kanazawa
  - Research Site, Kitaadachi-gun
  - Research Site, Kobe
  - Research Site, Kurashiki-shi
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Natori-shi
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sayama
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Takatsuki-shi
  - Research Site, Wakayama
  - Research Site, Yokohama
- Mexico (2):
  - Research Site, México
  - Research Site, Oaxaca City
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Groningen
- Russia (4):
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Yekaterinburg
- South Korea (9):
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Jinju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Ulsan
- Spain (4):
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Zaragoza
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Stockholm
- Taiwan (7):
  - Research Site, Changhua
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (10):
  - Research Site, Aberdeen
  - Research Site, Bristol
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Huddersfield
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Nottingham
  - Research Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Markovets A, Merino Vega D, Abbosh C, Quinn K, Chang K, Wienke S, Hartmaier R, Barrett JC, Hodgson D. Variability of Circulating Tumor DNA Levels in Plasma Samples From Patients With Advanced Non-Small-Cell Lung Cancer in the Absence of Treatment. JCO Precis Oncol. 2025 Oct;9:e2500287. doi: 10.1200/PO-25-00287. Epub 2025 Oct 30. PMID 41166679
- [Derived] Murat-Onana ML, Ramalingam SS, Janne PA, Gray JE, Ahn MJ, John T, Yatabe Y, Huang X, Rukazenkov Y, Javey M, Brown H, Li-Sucholeiki X. EGFR mutation testing across the osimertinib clinical program. Lung Cancer. 2025 Jun;204:108549. doi: 10.1016/j.lungcan.2025.108549. Epub 2025 Apr 18. PMID 40311309
- [Derived] King-Kallimanis BL, Bhatnagar V, Horodniceanu EG, Chen TY, Kluetz PG. Timing is everything: The importance of patient-reported outcome assessment frequency when characterizing symptomatic adverse events. Clin Trials. 2022 Jun;19(3):267-273. doi: 10.1177/17407745221093935. Epub 2022 May 15. PMID 35575012
- [Derived] Singh J, Bourke S, Dyer M, Devlin N, Longworth L. An Analysis of 5-Level Version of EQ-5D Adjusting for Treatment Switching: The Case of Patients With Epidermal Growth Factor Receptor T790M-Positive Nonsmall Cell Lung Cancer Treated With Osimertinib. Value Health. 2022 Jul;25(7):1205-1211. doi: 10.1016/j.jval.2022.01.022. Epub 2022 Apr 2. PMID 35379563
- [Derived] Papadimitrakopoulou VA, Mok TS, Han JY, Ahn MJ, Delmonte A, Ramalingam SS, Kim SW, Shepherd FA, Laskin J, He Y, Akamatsu H, Theelen WSME, Su WC, John T, Sebastian M, Mann H, Miranda M, Laus G, Rukazenkov Y, Wu YL. Osimertinib versus platinum-pemetrexed for patients with EGFR T790M advanced NSCLC and progression on a prior EGFR-tyrosine kinase inhibitor: AURA3 overall survival analysis. Ann Oncol. 2020 Nov;31(11):1536-1544. doi: 10.1016/j.annonc.2020.08.2100. Epub 2020 Aug 27. PMID 32861806
- [Derived] Papadimitrakopoulou VA, Han JY, Ahn MJ, Ramalingam SS, Delmonte A, Hsia TC, Laskin J, Kim SW, He Y, Tsai CM, Hida T, Maemondo M, Kato T, Jenkins S, Patel S, Huang X, Laus G, Markovets A, Thress KS, Wu YL, Mok T. Epidermal growth factor receptor mutation analysis in tissue and plasma from the AURA3 trial: Osimertinib versus platinum-pemetrexed for T790M mutation-positive advanced non-small cell lung cancer. Cancer. 2020 Jan 15;126(2):373-380. doi: 10.1002/cncr.32503. Epub 2019 Nov 26. PMID 31769875
- [Derived] Wu YL, Ahn MJ, Garassino MC, Han JY, Katakami N, Kim HR, Hodge R, Kaur P, Brown AP, Ghiorghiu D, Papadimitrakopoulou VA, Mok TSK. CNS Efficacy of Osimertinib in Patients With T790M-Positive Advanced Non-Small-Cell Lung Cancer: Data From a Randomized Phase III Trial (AURA3). J Clin Oncol. 2018 Sep 10;36(26):2702-2709. doi: 10.1200/JCO.2018.77.9363. Epub 2018 Jul 30. PMID 30059262
- [Derived] Lee CK, Novello S, Ryden A, Mann H, Mok T. Patient-Reported Symptoms and Impact of Treatment With Osimertinib Versus Chemotherapy in Advanced Non-Small-Cell Lung Cancer: The AURA3 Trial. J Clin Oncol. 2018 Jun 20;36(18):1853-1860. doi: 10.1200/JCO.2017.77.2293. Epub 2018 May 7. PMID 29733770
- [Derived] Akamatsu H, Katakami N, Okamoto I, Kato T, Kim YH, Imamura F, Shinkai M, Hodge RA, Uchida H, Hida T. Osimertinib in Japanese patients with EGFR T790M mutation-positive advanced non-small-cell lung cancer: AURA3 trial. Cancer Sci. 2018 Jun;109(6):1930-1938. doi: 10.1111/cas.13623. Epub 2018 May 31. PMID 29697876
- [Derived] Mok TS, Wu Y-L, Ahn M-J, Garassino MC, Kim HR, Ramalingam SS, Shepherd FA, He Y, Akamatsu H, Theelen WS, Lee CK, Sebastian M, Templeton A, Mann H, Marotti M, Ghiorghiu S, Papadimitrakopoulou VA; AURA3 Investigators. Osimertinib or Platinum-Pemetrexed in EGFR T790M-Positive Lung Cancer. N Engl J Med. 2017 Feb 16;376(7):629-640. doi: 10.1056/NEJMoa1612674. Epub 2016 Dec 6. PMID 27959700
- [Derived] Soria JC, Wu YL, Nakagawa K, Kim SW, Yang JJ, Ahn MJ, Wang J, Yang JC, Lu Y, Atagi S, Ponce S, Lee DH, Liu Y, Yoh K, Zhou JY, Shi X, Webster A, Jiang H, Mok TS. Gefitinib plus chemotherapy versus placebo plus chemotherapy in EGFR-mutation-positive non-small-cell lung cancer after progression on first-line gefitinib (IMPRESS): a phase 3 randomised trial. Lancet Oncol. 2015 Aug;16(8):990-8. doi: 10.1016/S1470-2045(15)00121-7. Epub 2015 Jul 6. PMID 26159065
- See also: D5160C00003AURA3_CSPredacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2892&filename=D5160C00003AURA3_CSPredacted.pdf
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00003&attachmentIdentifier=7ea80d41-31f4-44b2-8b95-0a1b2d616487&fileName=D5160C00003_SAP_ed4_redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00003&attachmentIdentifier=d5305855-1732-4dc0-bcfb-8c90e82a918f&fileName=d5160c00003-study-synopsis_DCO4_20Aug2019_-_Redactednew.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient dosed: 20 August 2014. Data cut off: 15 March 2019. Open for enrolment at 145 study centres, 126 centres in 17 countries randomised patients to treatment. Following the final OS analysis, patients were permitted to continue to receive treatment if, in the investigator's opinion, they were continuing to receive benefit from treatment. The last patient completed the study on the 15 December 2023
Groups:
- Osimertinib 80 mg: Daily single dose of Osimertinib 80mg
- Chemotherapy: Platinum-based doublet chemotherapy
Period: Overall Study
Arm/Group | Osimertinib 80 mg | Chemotherapy
Started | 279 | 140
Received Randomised Treatment Only | 279 | 136
Did Not Receive Treatment | 0 | 4
Crossed Over Osimertinib | 0 | 99 (Patients randomised to chemotherapy were allowed to crossover to Osimertinib after progression)
Completed | 60 | 27
Not Completed | 219 | 113
Not completed — Death | 184 | 88
Not completed — Lost to Follow-up | 7 | 1
Not completed — Withdrawal by Subject | 27 | 21
Not completed — Eligibility criteria not fulfilled | 0 | 1
Not completed — Other reasons | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Osimertinib 80 mg | Chemotherapy | Total
Number analyzed (Participants) | 279 | 140 | 419
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (11.64) [25 to 85] | 62.0 (11.91) [20 to 90] | 61.7 (11.72) [20 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 97 | 269
  Male | 107 | 43 | 150
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 182 | 92 | 274
  Black Or African American | 4 | 1 | 5
  Other | 4 | 1 | 5
  White | 89 | 45 | 134
  American Indian or Alaska Native | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by Investigator Assessment
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Progressive Disease (PD): >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of NTLs or a new lesion. PFS is the time from date of randomisation until the date of PD (by investigator assessment) or death (by any cause in the absence of progression) regardless of whether the patient withdrew from randomised therapy or received another anti-cancer therapy prior to progression. Patients who had not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST 1.1 assessment.
Time Frame: RECIST tumour assessments every 6 weeks from randomisation until objective disease progression up to 19 months (at the time of the primary PFS analysis).
Population: Full Analysis Set (All randomised patients)
Measure: Median (95% Confidence Interval); unit: Months
Units Other Than Participants: Events
Groups:
- Osimertinib 80mg: Daily single dose of Osimertinib 80mg
Arm/Group | Osimertinib 80mg | Chemotherapy
Number analyzed (Participants) | 279 | 140
Number analyzed (Events) | 140 | 110
Months | 10.1 [8.3 to 12.3] | 4.4 [4.2 to 5.6]
Statistical Analysis 1: Comparison: Osimertinib 80mg vs Chemotherapy; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.23 to 0.41] — A hazard ratio <1 favours Osimertinib 80mg

2. Secondary Outcome: Objective Response Rate (ORR) by Investigator Assessment
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. ORR is the percentage of patients with at least 1 visit response of CR or PR prior to progression or any further therapy.
Time Frame: as for outcome 1
Population: Full Analysis Set (All randomised patients)
Measure: Number; unit: % of participants
Arm/Group | Osimertinib 80mg | Chemotherapy
Number analyzed (Participants) | 279 | 140
% of participants | 70.6 | 31.4
Statistical Analysis 1: Comparison: Osimertinib 80mg vs Chemotherapy; Test type: Superiority or Other; p < 0.001, Regression, Logistic; adjusted for ethnicity (Asian/non-Asian); Odds Ratio (OR) = 5.39, 95% CI 2-sided [3.47 to 8.48] — odds ratio >1.0 favours Osimertinib 80 mg

3. Secondary Outcome: Duration of Response (DoR) by Investigator Assessment
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. DoR is the time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Time Frame: as for outcome 1
Population: Full Analysis Set (All randomised patients)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Osimertinib 80mg | Chemotherapy
Number analyzed (Participants) | 279 | 140
months | 9.7 [8.3 to 11.6] | 4.1 [3.0 to 5.6]
Statistical Analysis 1: Comparison: Osimertinib 80mg vs Chemotherapy; Test type: Superiority or Other; p < 0.001, formulae provided in Ellis S et al 2008; Treatments compared by calculating the ratio of the Expected (DoR) using the Log Normal probability distribution for DOR in responding patients; Ratio of Expected (DoR) = 6.22, 95% CI 2-sided [4.04 to 9.57]

4. Secondary Outcome: Disease Control Rate (DCR) by Investigator Assessment
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions; Stable disease (SD): Neither sufficient shrinkage to qualify as a response nor sufficient growth to qualify as progression; Progressive Disease (PD): >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of NTLs or a new lesion. DCR is the percentage of patients with best response of CR, PR or SD at >=6 weeks, prior to any progressive disease (PD).
Time Frame: as for outcome 1
Population: Full Analysis Set (All randomised patients)
Measure: Number; unit: % of participants
Arm/Group | Osimertinib 80mg | Chemotherapy
Number analyzed (Participants) | 279 | 140
% of participants | 93.2 [8.3 to 11.6] | 74.3 [3.0 to 5.6]
Statistical Analysis 1: Comparison: Osimertinib 80mg vs Chemotherapy; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.76, 95% CI 2-sided [2.64 to 8.84] — odds ratio >1.0 favours Osimertinib 80 mg

5. Secondary Outcome: Tumour Shrinkage by Investigator Assessment
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Tumour size was calculated as the sum of the longest diameters (SLD) of the Target Lesions. Tumour shrinkage is percentage change in tumour size from baseline using RECIST v1.1 tumour response.
Time Frame: as for outcome 1
Population: Full Analysis Set (All randomised patients)
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Osimertinib 80mg | Chemotherapy
Number analyzed (Participants) | 278 | 131
% change from baseline | -46.1 (29.50) | -24.4 (29.27)
Statistical Analysis 1: Comparison: Osimertinib 80mg vs Chemotherapy; Test type: Superiority or Other; p < 0.001, ANCOVA; Covariates for ethnicity (Asian, non-Asian) and the baseline sum of diameters of target lesions; Difference in LS means = -21.62, 95% CI 2-sided [-27.71 to -15.52] — LS Mean: Osimertinib -46.93, Chemo -25.3 A difference in LS means <0 favours Osimertinib 80mg

6. Secondary Outcome: Secondary: Overall Survival (OS)
Time Frame: From date of randomization until time of final OS analysis, a median follow-up of 43 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib 80mg | Chemotherapy
Number analyzed (Participants) | 279 | 140
Months | 26.8 [23.5 to 31.5] | 22.5 [20.2 to 28.8]
Statistical Analysis 1: Comparison: Osimertinib 80mg; Test type: Superiority or Other; p = 0.277, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.67 to 1.13] — A hazard ratio <1 favours Osimertinib 80 mg

7. Other Pre Specified Outcome: Time to First Subsequent Therapy (TFST)
Description: Time from randomisation to first subsequent anti-cancer therapy (FST) following randomised treatment discontinuation, or death if no FST administered. Any patient not known to have died nor received any subsequent anti-cancer therapy (ST) was censored at the last time known not to have received ST, ie, the last follow-up visit this was confirmed.
Time Frame: From date of randomisation until time of final OS analysis, a median follow-up of 43 months
Population: Full Analysis Set (All randomised patients)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib 80mg | Chemotherapy
Number analyzed (Participants) | 279 | 140
Months | 16.0 [13.8 to 18.4] | 6.0 [5.2 to 6.9]
Statistical Analysis 1: Comparison: Osimertinib 80mg vs Chemotherapy; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.16 to 0.28] — A hazard ratio <1 favors Osimertinib 80mg

8. Other Pre Specified Outcome: Time to Second Subsequent Therapy (TSST)
Description: Time from randomisation to second subsequent anti-cancer therapy (SST) following randomised treatment discontinuation, or death if no SST administered. Any patient not known to have died nor received any SST was censored at the last time known not to have received SST, ie, the last follow-up visit this was confirmed.
Time Frame: From date of randomisation until time of final OS analysis, a median follow-up of 43 months
Population: Full Analysis set (All randomised patients)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib 80mg | Chemotherapy
Number analyzed (Participants) | 279 | 140
Months | 20.0 [17.2 to 23.2] | 19.0 [16.5 to 22.0]
Statistical Analysis 1: Comparison: Osimertinib 80mg vs Chemotherapy; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.69 to 1.11] — A hazard ratio <1 favours Osimertinib 80 mg

ADVERSE EVENTS:
Time Frame: AEs from start of study drug until 28 days post treatment discontinuation up to 4 years and 7 months (at the time of analysis)
Description: Systematic assessment due to regular investigator assessment at study visits.
Arm/Group | Osimertinib 80 mg | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 188/279 | 93/136
Serious Adverse Events (participants affected / at risk) | 84/279 | 36/136
Other Adverse Events (participants affected / at risk) | 275/279 | 134/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osimertinib 80 mg (N=279) | Chemotherapy (N=136)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 3 (3)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 4 (4)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0)
Uterine cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
General physical health deterioratio (General disorders) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Organic brain syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Pharynx radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osimertinib 80 mg (N=279) | Chemotherapy (N=136)
Anaemia (Blood and lymphatic system disorders) | 32 (38) | 35 (45)
Leukopenia (Blood and lymphatic system disorders) | 14 (33) | 7 (12)
Neutropenia (Blood and lymphatic system disorders) | 14 (24) | 17 (26)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (30) | 10 (15)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 7 (7)
Lacrimation increased (Eye disorders) | 1 (1) | 8 (10)
Abdominal pain upper (Gastrointestinal disorders) | 10 (13) | 11 (11)
Constipation (Gastrointestinal disorders) | 50 (56) | 48 (94)
Diarrhoea (Gastrointestinal disorders) | 123 (226) | 14 (21)
Nausea (Gastrointestinal disorders) | 64 (75) | 66 (144)
Stomatitis (Gastrointestinal disorders) | 48 (70) | 22 (26)
Vomiting (Gastrointestinal disorders) | 42 (53) | 27 (49)
Asthenia (General disorders) | 23 (29) | 19 (25)
Fatigue (General disorders) | 54 (66) | 40 (60)
Malaise (General disorders) | 12 (14) | 14 (21)
Non-cardiac chest pain (General disorders) | 23 (24) | 6 (6)
Oedema peripheral (General disorders) | 16 (21) | 16 (23)
Pyrexia (General disorders) | 29 (36) | 13 (15)
Nasopharyngitis (Infections and infestations) | 34 (45) | 7 (7)
Paronychia (Infections and infestations) | 58 (72) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 36 (61) | 10 (10)
Urinary tract infection (Infections and infestations) | 24 (32) | 6 (9)
Alanine aminotransferase increased (Investigations) | 23 (34) | 17 (25)
Aspartate aminotransferase increased (Investigations) | 21 (33) | 16 (23)
Blood creatinine increased (Investigations) | 16 (20) | 9 (15)
Neutrophil count decreased (Investigations) | 17 (31) | 16 (38)
Platelet count decreased (Investigations) | 20 (32) | 21 (34)
Weight decreased (Investigations) | 16 (17) | 7 (7)
White blood cell count decreased (Investigations) | 22 (38) | 12 (36)
Decreased appetite (Metabolism and nutrition disorders) | 67 (78) | 49 (87)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (6) | 7 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (30) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 42 (52) | 14 (20)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 21 (25) | 8 (8)
Dizziness (Nervous system disorders) | 22 (26) | 12 (16)
Dysgeusia (Nervous system disorders) | 9 (9) | 12 (13)
Headache (Nervous system disorders) | 33 (44) | 16 (19)
Insomnia (Psychiatric disorders) | 26 (28) | 14 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 60 (72) | 20 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 35 (40) | 18 (20)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 41 (70) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 54 (66) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 42 (55) | 7 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 19 (25) | 3 (3)
Hypertension (Vascular disorders) | 9 (10) | 10 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (31) | 6 (11)
Abdominal pain (Gastrointestinal disorders) | 20 (22) | 6 (9)
Dyspepsia (Gastrointestinal disorders) | 15 (18) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 16 (26) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 (22) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 3 (3)
Skin fissures (Skin and subcutaneous tissue disorders) | 16 (18) | 1 (1)
Conjunctivitis (Infections and infestations) | 14 (17) | 5 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 21 (27) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review, should the submission for publication be delayed in order to file patent application. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT02151981/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT02151981/SAP_001.pdf